CLINICAL TRIAL: NCT04461782
Title: Interventional Study to Evaluate the Effect of a Food Supplement Comprising L. Plantarum After Oral Intake in Vaginal Microbiota
Brief Title: Interventional Study to Evaluate the Effect of the Oral Administration of L.Plantarum on Vaginal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AB-INTIMUS-Colonization
Record Dates: First submitted 2020-06-02; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Vaginal Infection
Keywords: vaginal probiotic
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactobacillus plantarum (Experimental): Oral intake 1 cap daily
  1E+09 cfu/cap of Lactobacillus plantarum
  Interventions: Dietary Supplement: Lactobacillus plantarum

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum — Oral food supplement

SUMMARY:
Vaginal microbiota is abundantly colonized by Lactobacillus genera. When vaginal microbiota gets altered, opportunistic microorganisms may proliferate and become abundant species giving rise to dysbiosis.

Probiotics are living organisms that provide the host certain benefits. Despite probiotics have been historically linked to intestinal microbiota, several research groups have published positive results for some Lactobacillus strains in vaginal microbiota. The Lactobacillus strain investigated in the presented project showed the ability to prevent recurrent vaginal Candidiasis in women with high vaginal candidiasis prevalence.

Nowadays the Lactobacillus strain here investigated is commercialized as vaginal caps, however oral intake is widely preferred among consumers. Because of that, this study aims to determine whether this Lactobacillus strain is able to colonize vaginal microbiota when administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects with vaginal microbiota classified as LBG (Lactobacillary grade) I, IIa or IIb.
* Using the same contraceptive within 4 weeks prior to study start.

Exclusion Criteria:

* Current vaginal infection.
* Vaginal infection 1 month prior to study start.
* Cervico-vaginal pathology.
* Papilloma human virus.
* Pregnant or breastfeeding mothers.
* Using IUD.
* Immunomodulators or systemic corticoids intake.
* Vaginal or systemic antibiotics intake 1 month prior to study start.
* Vaginal probiotic intake 1 month prior to study start.
* Less than three months after giving birth or abortion.
* Undergone vaginal or intestinal surgery three months prior to study start.
* Severe stress or depression.
* Systemic acute or severe disease.
* History of alcohol or drug abuse.
* Chronic intestinal pathology.
* Not understanding protocol procedures.
* Use of lubricant 24 hours or spermicide 7 days prior to study start.
* Swallowing difficulties.
* Impossibility to understand study procedures.
* Enrolled in another clinical study.
* Atrophic vaginitis not under treatment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Subjects must be female in order to sample vaginal microbiota
Enrollment: 30 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Colonization | change day 14-23 from baseline
  Determine the relative presence of Lactobacillus plantarum in vaginal microbiota by metagenomic analysis
Colonization | change day 42 from baseline
  Determine the relative presence of Lactobacillus plantarum in vaginal microbiota by metagenomic analysis

SECONDARY OUTCOMES:
Lactobacillary grade (LBG) score | change day 42 from baseline
  obtained by cytology analysis by pathologists and calculated according to Donders et al., 2002. Higher scores imply more severe conditions. Scale ranges from 1 to 3.
Other bacteria in vagina | change day 14-23 from baseline
  Detection of other bacteria by metagenomic analysis
Other bacteria in vagina | change day 42 from baseline
  Detection of other bacteria by metagenomic analysis
Vaginal pH | Change day 14-23 from baseline
  Measured through urine test strip
Vaginal pH | Change day 42 from baseline
  Measured through urine test strip
Product satisfaction | day 14-23
  Measured with a categorical scale (Likert type) going from 0 to 5 . Where 0 is very insatisfied and 5 is very satisfied
Safety and tolerability | through study completion, an average of 42 days
  Analyzed by the number of adverse events registered during the study
Gastrointestinal symptoms | Change day 14-23 from baseline
  Analyzed by the validated Spanish translation of Gastrointestinal Symptom Rating Scale (GSRS) according to Kulich et al., 2005. Score ranges from 0 to 90 where 0 is no symptoms at all and 90 is the highest severity in all symptoms assessed (e.g. pain, bloating, etc)

CONTACTS AND LOCATIONS:
Locations (1):
- Sta María del Rosell university hospital, Cartagena, Spain

REFERENCES:
- [Background] Reid G, Bruce AW. Urogenital infections in women: can probiotics help? Postgrad Med J. 2003 Aug;79(934):428-32. doi: 10.1136/pmj.79.934.428. PMID 12954951
- [Background] Guarner F, Schaafsma GJ. Probiotics. Int J Food Microbiol. 1998 Feb 17;39(3):237-8. doi: 10.1016/s0168-1605(97)00136-0. No abstract available. PMID 9553803
- [Background] Palacios S, Espadaler J, Fernandez-Moya JM, Prieto C, Salas N. Is it possible to prevent recurrent vulvovaginitis? The role of Lactobacillus plantarum I1001 (CECT7504). Eur J Clin Microbiol Infect Dis. 2016 Oct;35(10):1701-8. doi: 10.1007/s10096-016-2715-8. Epub 2016 Jul 9. PMID 27393491